CLINICAL TRIAL: NCT04216875
Title: Optimisation of Treatment of Chronic Patients With Diabetes Mellitus Type 2 in Primary Care (Qualiccare Begleitforschung Zur Optimierung Der Behandlung Von Chronischen Patienten Mit Diabetes Mellitus Typ 2 in Der Grundversorgung)
Brief Title: Best Practice Study of Diabetes Type 2 Management in Primary Care in Switzerland
Status: Completed | Type: Observational
Sponsor: QualiCCare (Other)
Collaborators: Swiss Society of Endocrinology and Diabetology (Unknown); Roche Diabetes Care (Industry); Sanofi (Industry); Concordia Versicherungen AG (Unknown); Novo Nordisk A/S (Industry); Galenica (Unknown)
Responsible Party: Sponsor
Other Study IDs: QualiCCare Diabetes III; BASEC Nr. 2017-01340 (Other: swissethics)
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Primary Care
Keywords: Best practice; optimisation of treatment; diabetes score; diabetes in primary care
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Primary Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- single primary care practices intervention: Independent primary care practices with one single medical doctor in the practice, usually ther owner of the practice working in his responsibility following the best practice procedure of the diabetes score.
  Interventions: Procedure: Best Practice Diabetes Management in Primary Care
- primary care group practice intervention: Independent primary care practices with more than one medical doctor working in their responsibility following the best practice procedure of the diabetes score.
  Interventions: Procedure: Best Practice Diabetes Management in Primary Care
- single primary care practices no intervention: Independent primary care practices with one single medical doctor in the practice, usually ther owner of the practice working in his responsibility without the intervention (not using Diabetes score)
- primary care group practice no intervention: Independent primary care practices with more than one medical doctor working in their responsibility without the intervention (not using Diabetes score).

INTERVENTIONS:
Procedure: Best Practice Diabetes Management in Primary Care — Practice adherence to best practice guidelines treating diabetes patients in different primary care practices is shown in this before- and after observational study
  Other Names: Diabetes Score
  Groups: primary care group practice intervention; single primary care practices intervention

SUMMARY:
This observational study intends to evaluate the use and adherence of different types of primary care practices to the diabetes criteria-protocol (diabetes score), developed by the Swiss Society of Endocrinology and Diabetology. This diabetes score comprises visits to the doctor, lifestyle consultations, clinical measures such as blood pressure, cholesterol or blood sugar, as well as measures concerning the prevention of secondary complications like kidney, eye or feet issues. The participating primary care practices need to treat 80% of their diabetes patients (their "diabetes population") in accordance to the score-criteria. In addition to the adherence to the eight score-criteria, the practices are required to also document statistically if their diabetes patients get the following medication: oral antidiabetics, insulin, blood pressure medication, statins and / flu vaccine. As this observational study is and before-and-after study, the primary care practices need to document for each of their diabetes patients the care they provided in the year before the introduction of the score-criteria and in the year following their introduction. Participating primary care practices ask their diabetes patients' consent to the documentation and anonymous transmittance of their data. Data evaluation is anonymous and on a population-based level (as opposed to individual-based). The hypothesis of the study is to prove that the implementation of evidence-based measures, such as a diabetes score can increase the treatment quality of diabetes patients in primary care practices and this increase is independent of the primary care practice structure in which it is applied.

DETAILED DESCRIPTION:
Information of the primary care practices regarding the background and goal of the project by means of a letter and informative documentation.

Recruitment of primary care practices, divided into three different practice organisations (individual practices and group practices run on a private basis and with financial autonomy, as well as forms of joint practices with employed physicians without financial autonomy).

A signed contract between QualiCCare and participating primary care practices regulates the collaboration.

Procedure:

A baseline documentation takes place retrospectively from the training/workshop for the past 12 months, and a second, prospective documentation of the treatment is done during the following 12 months.

Training of the participating general practioners (GP) and practice coordinator on the project including evaluation software, data entry and background to the criteria.

Documentation of the treatment quality of all patients with diabetes mellitus type 2 in a practice structure that meets the inclusion criteria according to the score criteria (baseline).

After 12 months, the treatment quality of the included patients with diabetes type 2 is recorded again using the same score.

ELIGIBILITY:
Inclusion Criteria:

* all patients in the primary care practice with a diabetes diagnosis, meaning their patient record shows that the patient either had an HbA1c value higher than 6.4 percent, takes insulin or oral antidiabetics and is treated at least during nine months in the participating primary care practice.

Exclusion Criteria:

* treatment in participating primary care practice during less than nine months (due to change of primary care provider, death, diabetes treatment solely by specialist);
* patients who do not give their patient consent to participate in study;
* patients whom the primary care provider excludes from study due to frailty, end of life or other reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population comprises two different kinds of primary care practices who either get the intervention or have no intervention (4 groups in total):
  single practices with one general practioner and group practices with several general practitioners. On the practice level, the study population comprises all diabetes patients who correspond to the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 738 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in score result before and after the introduction of the diabetes score criteria for treatment of diabetes patients in the primary care setting | one year
  The change is measured at baseline, before the introduction of the diabetes score criteria and one year after the introduction.
  There are 8 score criteria for the good diabetes management in primary care (such as 1x/y lifestyle consultation, 1x/foot control, etc). Each criteria gets a certain number of points if 80% of the participating patients are treated in accordance to the given criteria. In total, a maximum of 100 points can be achieved. The objective is to achieved a minimum of 70% (= 70 points).

SECONDARY OUTCOMES:
Evaluation of feasibility of the implementation of the diabetes score criteria in different primary care practice types | one year
  In order to test the feasibility of the use in different primary care practice types, the diabetes score criteria (as described above) are used in independent single practices and group practices. The above mentioned diabetes score consists of 8 score criteria concerning the diabetes management in primary care. The maximum amount of points are 100. it is desirable to achieve 70/100 points, whereas the points are attributed if 80% of the participating diabetes patients in the practice are treated according the the criteria.
Comparison of the diabetes treatment in regards to the different primary care settings | one year
  The resulting average score value of the diabetes treatment using the above described and mentioned diabetes score criteria in independent single primary care practices is compared with the resulting average score value of the diabetes treatment in group practices. The higher the score value, the better the treatment of diabetes patients in the respective practice structure (single or group practice).
Evaluation of practice tool used for the documentation and evaluation of the diabetes score | one year
  The participating primary care practices evaluate the practice tool and give feedback in regards to practicality and applicability in the respective practice setting

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Christ, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Hausarztmedizin KSSG, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christ E, Czock A, Renstrom F, Ammeter T, Ebrahimi F, Zechmann S, Kutz A, Diem P, Hauptle C, Brandle M. Evaluation of type 2 diabetes care management in nine primary care practices before and after implementation of the Criteria of Good Disease Management of Diabetes established by the Swiss Society of Endocrinology and Diabetology. Swiss Med Wkly. 2022 Jul 26;152:w30197. doi: 10.4414/smw.2022.w30197. eCollection 2022 Jul 18. PMID 35925612
- See also: official guideline platform of the Swiss medical Society FMH — https://www.guidelines.fmh.ch/index_detail.cfm?id=7B1EBC1C450FBB40A7CE5FA9B4DC4D6F

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study protocol and statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT04216875/Prot_SAP_ICF_000.pdf
  • Informed Consent Form: Informed Consent Form document (translated) (2017-09-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT04216875/ICF_001.pdf